CLINICAL TRIAL: NCT04820231
Title: The Effect of Platelet-Rich Plasma Injection on Pain, Function and Quality of Life in Patients With Hip Osteoarthritis
Brief Title: Platelet-Rich Plasma and Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Selda Çiftci, Specialist, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 191
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Hip Osteoarthritis
Keywords: hip osteoarthritis; platelet-rich plasma; ultrasound guidance
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: The patients with mono-lateral hip pain , grade 1 or 2 hip osteoarthritis according to the Kellgren-Lawrence classification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP injection group (Other): Intra-articular PRP injection with ultrasound guidance
  Three times PRP injections with an interval of one week
  Interventions: Other: intra-articular PRP injection

INTERVENTIONS:
Other: intra-articular PRP injection

SUMMARY:
To evaluate the effect of platelet-rich plasma (PRP) injection on pain, function and quality of life in patients with hip osteoarthritis.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent will undergo study entry.

Each patient received three times intra-articuler injections of PRP under ultrasound guidance, and they were administered once a week.

Baseline: Visual Analog Scale (VAS) including movement, rest and night, the Western Ontario and McMaster University Osteoarthritis Index (WOMAC) and SF-36 assessment

1st month: VAS, WOMAC and SF-36 assessment

3rd month: VAS, WOMAC and SF-36 assessment

6th month: VAS, WOMAC and SF-36 assessment

ELIGIBILITY:
Inclusion Criteria:

* Hip pain VAS > 4
* Grade 1 and 2 osteoarthritis according to the Kellgren-Lawrence classification
* No pathologies in the laboratory and coagulation parameters

Exclusion Criteria:

* Rheumatological disease with hip involvement
* Systemic active infection
* Severe cardiovascular disease
* Malignancy
* NSAID usage in the last week
* History of hip joint surgery
* History of traumatic hip injury
* Hgb values < 11 gr/dl
* Platelets values < 150.000 / µl
* History of bleeding disorder

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Visual Analog Scale (VAS) score at 1-month, 3-month and 6-month | Baseline, 1st month, 3rd month, 6th month
  The VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 'no pain' and 'worst pain'.
Change from baseline Western Ontario and McMaster University Osteoarthritis Index (WOMAC) score at 1-month, 3-month and 6-month | Baseline, 1st month, 3rd month, 6th month
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.
  Higher scores: worse pain, stiffness, and functional limitations.
Change from baseline SF-36 score at 1-month, 3-month and 6-month | Baseline, 1st month, 3rd month, 6th month
  The SF-36 is a 36-item self-report measure of health-related quality of life. It has eight subscales measuring different domains of health-related quality of life: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health . Two component scores are derived from the eight subscales: a physical health component score and a mental health component score.
  High scores: good quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jülide Öncü Alptekin, Study Chair — Şişli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Şişli, Turkey (Türkiye)